CLINICAL TRIAL: NCT00877812
Title: Vitamin B6 Dependence of One-Carbon Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01 D072398
Record Dates: First submitted 2009-04-01; First posted 2009-04-08 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Vitamin B6 Deficiency
Keywords: Vitamin B6; Vitamin B6 deficiency; Amino acids; pyridoxine
MeSH Terms: conditions — Vitamin B 6 Deficiency | interventions — Leucine; Amino Acids; Methionine; Serine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 glycine and leucine infusion (Experimental): Determine in healthy, adequately pyridoxine nourished humans using a protocol based on amino acid glycine tracer methods: (a) the postprandial rates of in vivo glycine turnover, glycine-based generation of one-carbon units, thymidylate and purine synthesis, and the impact of vitamin B6 deficiency on the rates of these processes and (b) the effect of vitamin B6 deficiency on the postprandial rate of glutathione synthesis. 14 subjects will be chosen after screening is complete and will begin a B6 deficient diet for 30 days. At the beginning and end of the 30 days they will receive an infusion of leucine and glycine then they will begin the four week diet. At the end of four weeks the infusion will be repeated.
  Interventions: Dietary Supplement: Arm 1 glycine and leucine
- Arm 2 Intervention of Serine and methionine infusion (Experimental): This arm will allow investigation of total Hcy remethylation and remethylation from serine-derived 1C units, kinetics of serine and the methionine cycle and kinetics of transsulfuration reactions. 14 healthy subjects will be selected and screened. Prior to starting a B6 deficient diet for four weeks an infusion of serine and methionine will commence. Following the first infusion the diet will begin and after four weeks another infusion will be done.
  Interventions: Dietary Supplement: Arm 2 Intervention of Serine and methionine infusion

INTERVENTIONS:
Dietary Supplement: Arm 1 glycine and leucine — Arm 1 glycine and leucine: A subset of 14 participants out of the total enrolled participants with an adequate nutritional status will undergo the tracer infusion of glycine and leucine amino acids protocol while an adequate vitamin pyridoxine, B6 status. After the first infusion each participant will then begin a diet low in vitamin B6 (<0.5 mg/d) for 4 weeks to achieve marginal B6 status followed by a repeat of fasting blood sampling and tracer infusion protocol.
  Other Names: amino acids; B6; leucine; methionine; deficieny
  Arms: Arm 1 glycine and leucine infusion
Dietary Supplement: Arm 2 Intervention of Serine and methionine infusion — Arm 2 Intervention of Serine and methionine infusion: A subset of 14 participants out of the total enrolled participants. Received an adequate nutritional status will undergo the tracer infusion of methionine and serine amino acids protocol while in adequate vitamin pyridoxine, B6 status. After the first infusion each subject will then begin a diet low in vitamin B6 (<0.5 mg/d) for 4 weeks to achieve marginal B6 status followed by repeat of fasting blood sampling and tracer infusion protocol.
  Other Names: B6 deficiency; methionine; serine
  Arms: Arm 2 Intervention of Serine and methionine infusion

SUMMARY:
Marginal vitamin B6 deficiency, which occurs commonly worldwide, leads to a cellular deficiency of the coenzyme pyridoxal phosphate (PLP). PLP is a coenzyme in several phases of one carbon (1C) metabolism, which is the array of reactions in which one carbon units are acquired and used in reactions including nucleotide synthesis, regeneration of methionine (Met) from homocysteine (Hcy), and methylation of many biological compounds. 1C metabolism is linked to the transsulfuration pathway in which Hcy undergoes PLP-dependent catabolism leading to cysteine, whose availability governs the formation of the antioxidant glutathione. Nutritional or genetic conditions that impair 1C metabolism are associated with elevation in plasma Hcy concentration and increased risk of vascular disease. It is believed that the metabolic effects of vitamin B6 deficiency will be most pronounced following protein intake when the vitamin B6-dependent pathways of amino acid metabolism experience the greatest substrate load. The human subjects protocols of this study consist of two distinct phases intended to extend our understanding of basic human 1C metabolism and the effects of marginal vitamin B6 deficiency under postprandial conditions. Phase 1 will investigate the effects of vitamin B6 nutrition on the PLP-dependent generation of 1C units by the glycine cleavage system and on the synthesis of glutathione. Phase 2 will investigate the dependence of methionine metabolism on vitamin B6 nutritional status, with particular emphasis on the recycling of Hcy to Met. Each phase of this study will involve 14 healthy, nutritionally adequate, young adults (7 male, 7 female) who will undergo metabolite profiling and kinetic analysis using intravenously infused stable isotopic tracers performed both before and after a ~4-week period of dietary vitamin B6 restriction. Subjects will be assigned to either Phase 1 or Phase 2, which will be identical in design except for the tracers and analytical methods used. We hypothesize that vitamin B6 deficiency will yield reduction in postprandial rates of homocysteine remethylation, generation of 1C units from glycine, and synthesis of glutathione. The results of this study will aid in assessing the consequences of nutritional and genetic variables affecting human metabolism and will further our understanding of the relationships between vitamin B6 nutrition and disease.

DETAILED DESCRIPTION:
If you volunteer for this study, you will come to the General Clinical Research Center (GCRC) at Shands Hospital for a screening visit. There approximately 27.5 mL of blood (5 1/2 teaspoons) will be taken from a vein in your arm. This will be used for tests to determine whether you are receiving adequate amounts of vitamin B6 and other vitamins, to analyze a part of the genetic information in certain blood cells that relates to how your body processes some nutrients, and to confirm your general health. If the vitamin B6 content of your blood is higher than the range needed for this study, which sometimes occurs from eating fortified foods, you might be asked to give another blood sample (2 teaspoons) after several weeks to have the screening test repeated. You will also be asked questions about your health and a detailed assessment of your regular diet will be carried out. Your general health will be confirmed by taking a medical history, physical exam, and standard blood tests including liver, kidney, bone marrow function, cholesterol and urine analysis. To take part in this study, you must be in good health and in adequate nutritional status for vitamin B6 and other vitamins.

Because of risks to a developing fetus from inadequate vitamin B6 intake, a pregnancy test will be conducted with females three times during the study (during the screening visit and before each hospital admission) and women who participate in this study should use protection to prevent pregnancy during the study; if you become pregnant you will be released from the study.

Once you have completed all screening procedures you will be asked to eat meals prepared by the GCRC for 2 days, you will then participate in the procedure to test how effectively vitamin B6 functions in helping your body use certain amino acids. This will involve giving you a solution of certain amino acids by a vein in your arm over the course of 9 hours.

On the evening before this procedure, you will report to the GCRC at approximately 8:00 p.m. You will spend the night at the GCRC and will not be allowed to eat after 9:00 p.m. On the following morning, you will not be given breakfast. You will have an intravenous catheter placed into a vein in each arm, one for blood samples to be taken throughout the day, and one for the amino acid solution to be given. You will also be asked to breath (one breath) through a straw into a glass tube at different times, while the amino acid solution is being given. Before starting the amino acid solution, a blood sample (about 7 teaspoons) will be taken from a vein in one arm. Then the solution containing amino acids and nucleotides will be pumped slowly into your blood over the next 9-hour period. You will not be allowed to eat normal foods during this 9-hour period. However, you will be given a liquid nutritional formula to drink each hour during the day (starting after the first blood sample is taken). Approximately 14 blood samples (9 mL, less than 2 teaspoons each) and 8 breath samples will be taken from you while you receive the amino acid solution. In addition, at 6 times during the day you will be asked to lie quietly for 10 minutes while breathing into a special, clear hood that will measure your metabolic rate (the rate at which your body uses energy). You will remain at the GCRC for the entire 9-hour period, although you will be able to do limited activities (TV and reading). At the end of the 9-hour period, you will be able to go home and resume your activities. The following day you will resume eating meals prepared by the GCRC. While at the GCRC on days 3 and 4 after this procedure, you will be asked to give two more blood samples, one in the morning and one in the evening, and on day 5 you will be asked to give one blood sample in the morning (2 teaspoons each).

The day after you are discharged from the GCRC, you will be asked to eat, for a period of approximately 4 weeks, a diet containing reduced amounts of vitamin B6 and limit the amount of caffeine (in coffee, tea, and carbonated drinks) you drink to one to two per day. Twice each day during this approximately 4 week period you will come to the General Clinical Research Center (GCRC) at Shands Hospital where you will eat your breakfast and evening meals. Also, you will be weighed once daily and have your heart rate, respirations and blood pressure monitored twice weekly. You will be given a sack lunch to be consumed wherever you choose. To be sure that you are getting adequate amounts of all nutrients except the vitamin being studied, you will be given a pill containing a vitamin and mineral supplement each day. Once each week (when you come into the GCRC to eat breakfast), you will have two teaspoons of blood taken from a vein in your arm to allow monitoring of your vitamin B6 status.

After finishing approximately 4 weeks on this diet, you will participate again in the procedure to test how effectively vitamin B6 functions in helping your body use certain amino acids. Again, this will involve giving you a solution of certain amino acids by a vein in your arm over the course of 9 hours. As before, you will report to the GCRC at approximately 8:00 p.m. on the evening before the procedure. You will spend the night at the GCRC and will not be allowed to eat after 9:00 p.m. The exact same procedures will be carried out as in the first admission.

A few days prior to the second admission, while you are on the GCRC receiving your diet, you will have the same general health blood and urine tests collected as you had done before the first admission.

When the amino acid solution has been completely given, approximately 9 hours, you will be able to go home and resume your activities. You will be asked to return to the GCRC to give blood samples on days 3, 4, and 5 after this procedure just as you did after the first admission. You will then be finished with the study. You will be given a 30 day supply of vitamin and mineral supplements to be taken daily to be sure that your body gets adequate amounts of vitamin B6 and other nutrients.

After the laboratory analysis of blood samples from this study has been completed, if you agree, some of the samples will be kept in frozen storage for possible future analysis of nutrients or genetic information related to how your body processes nutrients. Please refer to the Addendum for Blood Storage and Future Testing attached.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years of age
* adequate vitamin B6 levels
* not pregnant

Exclusion Criteria:

* abnormal labs
* pregnancy
* on medications

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Hypothesis Aim 1 | One year
  (a) Vitamin B6 deficiency will reduce the rate of glycine turnover and interconversion with serine and will reduce the generation of 1C units by the glycine cleavage system. (b) Vitamin B6 deficiency will yield a reduced in vivo rate of erythrocyte glutathione synthesis.
Hypotheses Aim 2 | 30 days
  (a) Vitamin B6 deficiency will reduce the in vivo rate of generation of one-carbon units from serine and, thus, overall homocysteine remethylation. (b) In vivo rates of cysteine synthesis will be reduced in vitamin B6 deficiency. (c) Thymidylate synthesis from serine-derived one-carbon units will be reduced during vitamin B6 deficiency

SECONDARY OUTCOMES:
Hypotheses Aim 3 | 30 days
  (a) Vitamin B6 deficiency will yield increased plasma glycine, cystathionine and glutathione but decreased erythrocyte glutathione concentration. (b) Vitamin B6 deficiency will cause reduced activity of lymphocyte SHMT and the glycine cleavage system and reduced cellular (lymphocyte) glycine concentration..

CONTACTS AND LOCATIONS:
Overall Officials: Jesse F Gregory, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Lamers Y, Williamson J, Gilbert LR, Stacpoole PW, Gregory JF 3rd. Glycine turnover and decarboxylation rate quantified in healthy men and women using primed, constant infusions of [1,2-(13)C2]glycine and [(2)H3]leucine. J Nutr. 2007 Dec;137(12):2647-52. doi: 10.1093/jn/137.12.2647. PMID 18029478
- [Result] Lamers Y, Coats B, Ralat M, Quinlivan EP, Stacpoole PW, Gregory JF 3rd. Moderate vitamin B-6 restriction does not alter postprandial methionine cycle rates of remethylation, transmethylation, and total transsulfuration but increases the fractional synthesis rate of cystathionine in healthy young men and women. J Nutr. 2011 May;141(5):835-42. doi: 10.3945/jn.110.134197. Epub 2011 Mar 23. PMID 21430249
- [Result] Lamers Y, O'Rourke B, Gilbert LR, Keeling C, Matthews DE, Stacpoole PW, Gregory JF 3rd. Vitamin B-6 restriction tends to reduce the red blood cell glutathione synthesis rate without affecting red blood cell or plasma glutathione concentrations in healthy men and women. Am J Clin Nutr. 2009 Aug;90(2):336-43. doi: 10.3945/ajcn.2009.27747. Epub 2009 Jun 10. PMID 19515736
- [Result] Lamers Y, Williamson J, Ralat M, Quinlivan EP, Gilbert LR, Keeling C, Stevens RD, Newgard CB, Ueland PM, Meyer K, Fredriksen A, Stacpoole PW, Gregory JF 3rd. Moderate dietary vitamin B-6 restriction raises plasma glycine and cystathionine concentrations while minimally affecting the rates of glycine turnover and glycine cleavage in healthy men and women. J Nutr. 2009 Mar;139(3):452-60. doi: 10.3945/jn.108.099184. Epub 2009 Jan 21. PMID 19158217
- [Derived] DeRatt BN, Ralat MA, Gregory JF. Short-Term Vitamin B-6 Restriction Does Not Affect Plasma Concentrations of Hydrogen Sulfide Biomarkers Lanthionine and Homolanthionine in Healthy Men and Women. J Nutr. 2015 Apr 1;146(4):714-719. doi: 10.3945/jn.115.227819. PMID 26962179
- [Derived] Gregory JF, DeRatt BN, Rios-Avila L, Ralat M, Stacpoole PW. Vitamin B6 nutritional status and cellular availability of pyridoxal 5'-phosphate govern the function of the transsulfuration pathway's canonical reactions and hydrogen sulfide production via side reactions. Biochimie. 2016 Jul;126:21-6. doi: 10.1016/j.biochi.2015.12.020. Epub 2016 Jan 4. PMID 26765812
- [Derived] Rios-Avila L, Coats B, Chi YY, Midttun O, Ueland PM, Stacpoole PW, Gregory JF 3rd. Metabolite profile analysis reveals association of vitamin B-6 with metabolites related to one-carbon metabolism and tryptophan catabolism but not with biomarkers of inflammation in oral contraceptive users and reveals the effects of oral contraceptives on these processes. J Nutr. 2015 Jan;145(1):87-95. doi: 10.3945/jn.114.201095. Epub 2014 Nov 19. PMID 25527663